CLINICAL TRIAL: NCT04764903
Title: A Retrospective Review of the Association of Baseline Characteristics of Male Patients Presented With Lower Urinary Tract and Long Term Clinical Outcomes
Brief Title: The Association of Baseline Characteristics of Male Patients Presented With LUTS and Long Term Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Fai NG, Professor, Chinese University of Hong Kong
Other Study IDs: CRE-2019.400
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LUTS/Nocturia: Patients with LUTS / Nocturia
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention in this study

SUMMARY:
Non-neurogenic male lower urinary tract symptom (LUTS) is one of the most common symptom presented in urological clinic. Male LUTS could be a result of a combination of many different conditions, including benign prostate hypertrophy, overactive bladder, diabetes, noctural polyuria, sleep apnoea etc. Also male LUTS has shown to have close relationship with metabolic and cardiovascular conditions. Because of the increasing evidences to suggest a close relationship of cardiovascular condition and metabolic problems and male LUTS, this is a study to retrospective review of the patients assessed in this urology clinic and have a more in-depth assessment of the relationship of the baseline characteristics of these medical conditions with the presenting symptoms, as well as the long term urological and overall clinical outcomes of these patients.

DETAILED DESCRIPTION:
This is a retrospective study.Male patients who presented with lower urinary tract symptom to our centre and assessed in the urology clinic from 2005 to 2019 would be enrolled to the study. This study will be conducted by observation; that is, data will be captured from medical records and central medical system (CMS), but patients will not be contacted. All the demographic and medical background, as well as investigations performed during the assessment including uroflowmetry, post-voiding residual, questionnaires, blood pressure, pulse, vascular assessment and blood result will be collected. Follow-up data including usage of medication, clinical outcomes (such as development of urinary retention, cardiovascular events, need of surgical intervention, mortality etc.) will be captured from the medical records.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 35 and 90 years old with LUTS/nocturia and received assessment at urology centre.

Exclusion Criteria:

* Men having history of prostatic surgery, prostate cancer, active urinary tract infection, aortic aneurysm, marked cardiac arrhythmia and severe peripheral vascular disease

Ages: 35 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: Male patients who presented with lower urinary tract symptom to our centre and assessed in the nurse-led pre-assessment clinic
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
The overall prevalence of adverse cardiovascular events (MACE) in male patients presented with lower urinary tract symptoms (LUTS) | Through study completion, an average of 2 years
  Major adverse cardiovascular events such as myocardial infraction, ischemic heart disease, heart failure, coronary angioplasty etc. in male patients with LUTS. It is assessed by medical record
The overall prevalence of diabetes in male patients presented with lower urinary tract symptoms (LUTS) | Through study completion, an average of 2 years
  It is assessed by medical record
The overall prevalence of dyslipidaemia in male patients presented with lower urinary tract symptoms (LUTS) | Through study completion, an average of 2 years
  It is assessed by medical record

SECONDARY OUTCOMES:
Correlation between nocturia and Central arterial stiffness (CAS) | Baseline
  Nocturia is assessed by International Prostate Symptom Score Question 7, high value means worser nocturia; CAS is assessed by brachial-ankle PWV (baPWV), the value >1800cm/sec is highly associated with development of MACE
Incidence of acute retention of urine | Through study completion, an average of 2 years
  It is assessed by medical record
Incidence of requirement of surgical intervention | Through study completion, an average of 2 years
  It is assessed by medical record
Overall mortality | Through study completion, an average of 2 years
  It is assessed by medical record

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

REFERENCES:
- [Background] Ng CF, Wong A, Li ML, Chan SY, Mak SK, Wong WS. The prevalence of cardiovascular risk factors in male patients who have lower urinary tract symptoms. Hong Kong Med J. 2007 Dec;13(6):421-6. PMID 18057428
- [Background] Yee CH, Yip JSY, Cheng NMY, Kwan CH, Li KM, Teoh JYC, Chiu PKF, Wong JH, Chan ESY, Chan CK, Hou SSM, Ng CF. The cardiovascular risk factors in men with lower urinary tract symptoms. World J Urol. 2019 Apr;37(4):727-733. doi: 10.1007/s00345-018-2432-2. Epub 2018 Aug 6. PMID 30083830
- [Background] Teoh JY, Chan CK, Wang MH, Leung CH, Chan ES, Chiu PK, Yee CH, Wong HM, Hou SS, Ng CF. Transurethral resection of prostate for acute urinary retention is linked to shorter survival in younger men. Asian J Androl. 2019 Sep-Oct;21(5):468-472. doi: 10.4103/aja.aja_101_18. PMID 30648670
- [Background] Everaert K, Anderson P, Wood R, Andersson FL, Holm-Larsen T. Nocturia is more bothersome than daytime LUTS: Results from an Observational, Real-life Practice Database including 8659 European and American LUTS patients. Int J Clin Pract. 2018 Jun;72(6):e13091. doi: 10.1111/ijcp.13091. Epub 2018 May 16. PMID 29767479